CLINICAL TRIAL: NCT00749151
Title: A Randomized Controlled Trial on the Effectiveness of the American Lung Association Reactive Anti-Smoking Telephone Help Line in Illinois
Brief Title: Effectiveness of the American Lung Association Reactive Anti-Smoking Telephone Help Line in Illinois
Acronym: QUITLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Akshay Sood, M.D., M.P.H., SIU School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SIUSOM-08-004
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Smoking
Keywords: smoking cessation; telephone help line
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Literature (No Intervention)
- Lit + Counseling (Experimental)
  Interventions: Behavioral: telephone counseling

INTERVENTIONS:
Behavioral: telephone counseling — First time callers to telephone help line agreed to one year follow-up on smoking cessation.
  Other Names: American Lung Association Quit Line
  Arms: Lit + Counseling

SUMMARY:
An estimated 47 million adult Americans smoke. The American Lung Association has launched a reactive telephone help line to assist in smoking cessation. The proposed study will evaluate its effectiveness in a randomized controlled trial design involving active smokers who call this helpline. Eligible callers will be randomized into two groups: those who receive self-help literature only (i.e. control group) and those who receive additional reactive telephone counseling (i.e. study group). Detailed information will be collected proactively by an independent research calling specialist from all subjects who enroll into the study, by way of follow-up telephone calls, at one, three, six and twelve months following the screen date. The outcome measures to be compared are abstinence rates, quit attempts, changes in extent of smoking and behavioral stage, and cost-effectiveness. A thousand subjects will be enrolled in the two study arms in equal numbers over a period of fifteen months. Intent to treat analysis will be used after adjustment for covariates. The significance of this study lies in establishing the public health importance of such a reactive telephone helpline as a low intensity and low cost interventional smoking cessation tool.

DETAILED DESCRIPTION:
An estimated 47 million adult Americans smoke. Telephone counseling is considered a promising mode of intervention for smoking cessation. While pro-active (acting in anticipation of future change) telephone counseling has been shown to be efficacious in randomized trials, evaluation of reactive (occurring as a result of a stimulus) phone lines has been criticized by the lack of randomization and adequate controls for comparison. The American Lung Association has launched a reactive telephone help line to assist in smoking cessation. The proposed study will evaluate its effectiveness in a randomized controlled trial design involving active smokers who call this helpline. Eligible callers will be randomized into two groups: those who receive self-help literature only (i.e. control group) and those who receive additional reactive telephone counseling (i.e. study group). Detailed information will be collected proactively by an independent research calling specialist from all subjects who enroll into the study, by way of follow-up telephone calls, at one, three, six and twelve months following the screen date. The outcome measures to be compared are abstinence rates, quit attempts, changes in extent of smoking and behavioral stage, and cost-effectiveness. A thousand subjects will be enrolled in the two study arms in equal numbers over a period of fifteen months. Intent to treat analysis will be used after adjustment for covariates. The significance of this study lies in establishing the public health importance of such a reactive telephone helpline as a low intensity and low cost interventional smoking cessation tool.

ELIGIBILITY:
Inclusion Criteria:

* Be an active nicotine user at the time of initial contact with the Tobacco
* Quitline, and interested in quitting nicotine
* Establish contact, by himself or herself, with the ALA, seeking help in quitting nicotine;
* Be contactable by telephone, and
* Be agreeable to consenting for the study and for follow-up by telephone interviews for a total period of six months

Exclusion Criteria:

* Pregnant subjects,
* Minors (under 18 years of age),
* People with current psychiatric conditions other than anxiety or depression,
* Refusal or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2002-12; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
point prevalence abstinence rate | not a single puff for 7 day minimum
continuous abstinence rate | calculated at 1, 3, and 6 months
change in behavioral stage with respect to smoking (transtheoretical model) | baseline, 1, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sood, MD, MPH, Principal Investigator — SIU School of Medicine
Locations (1):
- SIU School of Medicine, Springfield, Illinois, United States